CLINICAL TRIAL: NCT01492127
Title: Evolution of Plasma Proteasome Levels Following Curative Treatment of Hepatocellular Carcinoma in Cirrhotic Patients
Brief Title: Evaluation of Proteasome as a Marker of Hepatocellular Carcinoma in Cirrhotic Patients Following Curative Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UF 8671
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis
Keywords: Hepatocellular carcinoma; cirrhosis; proteasome; alpha-fetoprotein
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood test (No Intervention): Blood test :carcinoma in cirrhotic patients
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — Blood test

SUMMARY:
This study will evaluate the usefulness of plasma proteasome levels as a tumor marker of hepatocellular carcinoma (HCC) by studying their variation following curative treatment of HCC. The hypothesis of the study is that plasma proteasome levels will decrease following curative treatment, and that proteasome levels could be used as a marker to detect early recurrence.

DETAILED DESCRIPTION:
HCC occurs in the vast majority of cases in the context of cirrhosis. Cirrhosis is considered a pre-cancerous state, which justifies systematic screening for HCC. Screening currently relies on measurement of alpha-foetoprotein (AFP) levels and ultrasound scans every 4 to 6 months. However, AFP has poor sensitivity as a marker for HCC. We have recently shown that plasma proteasome levels have a higher sensitivity than HCC for detecting HCC in cirrhotic patients, particularly when the tumors are small and can still benefit from curative treatment. The hypothesis of the study is that plasma proteasome levels will decrease following curative treatment, and that proteasome levels could be used as a marker to detect early recurrence. The goal of this study is to determine whether plasma proteasome levels in cirrhotic patients with HCC decrease following curative treatment (radiofrequency, surgical resection, liver transplantation). Plasma proteasome levels will be measured before treatment and 3 months after treatment, then subsequently at 3 month intervals over one year following treatment. The variation of proteasome levels will be compared to AFP levels. The sensitivity of proteasome as a marker to detect tumor recurrence will be evaluated, and compared to AFP.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients with hepatocellular carcinoma proven by histological examination of a biopsy specimen, eligible for curative treatment (radiofrequency, surgical resection, liver transplantation)
* Patient able to give informed consent
* Patient with Social Security coverage

Exclusion Criteria:

* Secondary liver tumors
* Non hepatocellular carcinoma primary liver tumor
* Hepatocellular carcinoma without cirrhosis
* Patients with hepatocellular carcinoma and cirrhosis not eligible for curative treatment
* Prisoners
* Adults under guardianship or curatorship
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Variation of plasma proteasome | 3 months afterwards
  Variation of plasma proteasome levels before curative treatment of HCC and 3 months afterwards

SECONDARY OUTCOMES:
Variation of plasma proteasome | 6, 9 and 12 months
  Variation of plasma proteasome levels 6, 9 and 12 months following curative treatment for HCC, comparison with AFP levels and results from imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Funakoshi, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

REFERENCES:
- [Background] Henry L, Lavabre-Bertrand T, Vercambre L, Ramos J, Carillo S, Guiraud I, Pouderoux P, Bismuth M, Valats JC, Demattei C, Duny Y, Chaze I, Funakoshi N, Bureau JP, Daures JP, Blanc P. Plasma proteasome level is a reliable early marker of malignant transformation of liver cirrhosis. Gut. 2009 Jun;58(6):833-8. doi: 10.1136/gut.2008.157016. Epub 2009 Feb 6. PMID 19201777